CLINICAL TRIAL: NCT03646448
Title: Intervening in Problematic Internet Use - Preventive Measures for Risk Groups
Brief Title: Intervening in Problematic Internet Use
Acronym: iPIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government)
Responsible Party: Principal Investigator, Hans-Jürgen Rumpf, Head of Research group S:TEP, University of Luebeck
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1504/68405
Record Dates: First submitted 2018-03-20; First posted 2018-08-24 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Internet Use Disorders
Keywords: Internet Use Disorders; Brief Intervention; Motivational Interviewing; CBT; Proactive
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Counseling based on Motivational Interviewing and elements of Cognitive Behavioral Therapy
  Interventions: Behavioral: Motivational Interviewing
- Control group (No Intervention): Control group receiving a booklet on problematic Internet use

INTERVENTIONS:
Behavioral: Motivational Interviewing — Up to three counseling sessions on telephone based on Motivational Interviewing and elements of Cognitive Behavioral Therapy. Counselings are within 12 weeks after the baseline diagnostic interview and follow the stepped care approach.
  Arms: Intervention group

SUMMARY:
The present study examines the efficacy of a brief intervention for problematic Internet use based on Motivational Interviewing (MI) and Cognitive Behavioral Therapy (CBT) in a sample of students screened proactively in vocational schools in Northern Germany. Participants will be randomized in an intervention and a control group. It is hypothesized that after 12 months, participants of the intervention group fulfill less DSM-5 criteria for Internet use disorders, spend less time in the Internet, and suffer from less negative consequences caused by the problematic Internet use, compared to the control group.

DETAILED DESCRIPTION:
Problematic Internet use is an increasing problem, especially in younger age groups. A population-based study revealed elevated prevalences in adolescents and young adults. The present study aims to provide an intervention for this vulnerable group to change the problematic Internet use. This is suggested to prevent the development of more severe forms of dependence. Brief interventions using MI and elements of CBT have shown to be an adequate method to change addictive behaviors.

For the recruitment, students of vocational schools in the states of Schleswig-Holstein and Hamburg in Northern Germany are screened proactively in classes. Participants fulfilling at least 21 points on the Compulsive Internet Use Scale (CIUS) receive a diagnostic telephone interview. If fulfilling at least 2 DSM-5 criteria, participants will be randomly allocated to two conditions: (1) Intervention group with up to three telephone counseling sessions based on MI, (2) Control group receiving a booklet on problematic Internet use. Outcome measures are a reduction of DSM-5 criteria for Internet use disorders, a reduction of time spent on the Internet, and a reduction of negative consequences caused by the problematic Internet use. The efficacy of the intervention will be examined after 6 and 12 months in follow-up interviews.

ELIGIBILITY:
Inclusion Criteria:

* CIUS score of 21 and at least 2 DSM-criteria
* At least 16 years old

Exclusion Criteria:

* Current treatment for mental disorders

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 470 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Change of DSM-5 criteria | Assessment of criteria at baseline and at 6- and 12-month follow ups
  Criteria for Internet Use Disorders according to the Internet Gaming Disorder in the DSM-5, but for all Internet Applications are assessed with a diagnostic clinical interview based on the Composite International Diagnostic Interview (CIDI)
Change of time spent on the Internet | Assessment of time on the Internet at baseline and at 6- and 12-month follow ups
  Average time of private Internet use on a weekday and on weekends and maximum use are assessed at baseline and at 6- and 12-month follow ups. Change of time is measured by the difference between the follow up assessments and the baseline.
Change of disabilities caused by the problematic Internet use | Assessment of disabilities at baseline and at 6- and 12-month follow ups
  World Health Organization Disability Assessment Schedule 2.0 (WHODAS) 2.0 (Adapted Version for problematic Internet use):
  * 4 items ranging from 0 (no impairment) to 10 (strong impairment)
  * 2 items estimating the days of impairment in the past 12 months (time frame will be adapted to the time frame in the assessment)
  * For change of disabilities, the difference between follow up assessments and baseline will be measured for the single items.
Change of negative consequences caused by the problematic Internet use | Assessment of negative consequences at baseline and at 6- and 12-month follow ups
  Negative Consequences-Questionnaire from the Criminological Research Institute of Lower Saxony:
  * 8 items ranging from 1 (much worse) to 5 (much better)
  * Maximum sum score ranges from 8 to 40
  * The questionnaire is inversely coded, so higher outcomes provide a better outcome
  * For change of negative consequences, the difference between the sum scores in the follow up assessments and baseline will be measured

SECONDARY OUTCOMES:
Readiness to change Internet use | Assessment of readiness to change at baseline and at 6- and 12-month follow ups
  Readiness to change is measured with a single item ("How important would it be for you to change your Internet use behavior?") on a 10-point-Likert scale (1=not important at all, 10=very important). A higher value represents a better outcome.
Self-efficacy to change Internet use | Assessment of self-efficacy at baseline and at 6- and 12-month follow ups
  Self-efficacy is measured with a single item ("How confident are you to change your Internet use behavior?") on a 10-point-Likert scale (1=not confident at all, 10=very confident). A higher value represents a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Jürgen Rumpf, PD Dr., Principal Investigator — University of Lübeck
Locations (1):
- University of Lübeck, Lübeck, Germany